CLINICAL TRIAL: NCT01683604
Title: A Multi-National, Multi-Center Non-Interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab (ACT-UP)
Brief Title: Observational Study of Tocilizumab in Participants With Rheumatoid Arthritis in Australia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28144
Record Dates: First submitted 2012-09-05; First posted 2012-09-12 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis (RA) Participants (All Groups): Participants with severe RA were prescribed with tocilizumab in accordance with routine clinic practice, and were observed for 6 months.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
This multi-center, observational study will evaluate the treatment patterns in clinical practice, efficacy and safety of tocilizumab in participants with rheumatoid arthritis (RA) who have had an inadequate response (or were intolerant to) treatment with non-biological disease-modifying anti-rheumatic drugs (DMARDs) or with one biological agent. Data will be collected from each eligible participant initiated on tocilizumab treatment by their treating physician according to approved label for 6 months from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Severe RA.
* Inadequate response (or intolerant) to non-biological DMARDs or one biologic agent
* Participants initiating treatment with tocilizumab on their physician's decision (in accordance with the local label), including participants who started treatment with tocilizumab within the 8 weeks prior to the enrolment visit.

Exclusion Criteria:

* Tocilizumab treatment more than 8 weeks prior to the enrolment visit.
* Previous tocilizumab treatment in a clinical trial or for compassionate use.
* Enrolled in an ongoing clinical trial and/or treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with tocilizumab.
* History of autoimmune disease or any joint inflammatory disease other than RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA participants treated with tocilizumab
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Australia (7):
  - Campsie, New South Wales
  - Coffs Harbour, New South Wales
  - New Lambton, New South Wales
  - Woodville, South Australia
  - Heidelberg, Victoria
  - Morwell, Victoria
  - Shenton Park, Western Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis (RA) Participants (All Groups): Participants with severe RA were prescribed with tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) Participants (All Groups)
Started | 37
Completed | 32
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled participants who received at least 1 dose of tocilizumab.
Groups:
- RA Participants (All Groups): Participants with severe RA were prescribed with tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
Arm/Group | RA Participants (All Groups)
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab Treatment at Month 6 After Treatment Initiation
Description: Percentage of participants on tocilizumab treatment at Month 6 was calculated as: [(participants on tocilizumab treatment at Month 6) divided by (participants evaluable for primary objective)] multiplied by 100.
Time Frame: Month 6
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- RA Participants (Biologic Naïve Group): Participants with severe RA, and no prior exposure to biologic agent were prescribed with tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
- RA Participants (Biologic Exposed Group): Participants with severe RA, with prior exposure to biologic agent were prescribed with tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
- RA Participants (Monotherapy Group): Participants with severe RA, were prescribed with tocilizumab alone, in accordance with routine clinic practice and were observed for 6 months.
- RA Participants (Combination Therapy Group): Participants with severe RA, were prescribed with disease-modifying anti-rheumatic drug (DMARD) at the time of first dose of tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
percentage of participants | 79.3 | 100 | 80 | 84.4 | 83.8

2. Primary Outcome: Patient Assessment of Pain Using Visual Analog Scale (VAS) at Baseline
Description: Participants measured the pain intensity due to RA on a 100 millimeter (mm) VAS, where the responses were on a continuous range from 0 = no pain to 100 = unbearable pain.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Groups:
- RA Participants (Combination Therapy Group): Participants with severe RA, were prescribed with DMARD at the time of first dose of tocilizumab, in accordance with routine clinic practice and were observed for 6 months.
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
millimeters (mm) | 60.1 (31.08) | 47.2 (31.93) | 79.3 (19.55) | 55.3 (31.49) | 57.6 (31.14)

3. Primary Outcome: Patient Global Assessment of Disease Activity Using VAS at Baseline
Description: The patient's global assessment of disease activity was measured using a 100 mm VAS, where the responses were on a continuous range from 0 = managing very well to 100 = managing very poorly.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 24 | 6 | 3 | 27 | 30
mm | 69.6 (29.71) | 59.0 (33.03) | 85.0 (11.36) | 65.5 (31.02) | 67.5 (30.11)

4. Primary Outcome: Physician Global Assessment of Disease Activity Using VAS at Baseline
Description: Physician global assessment of disease activity was assessed on a 100 mm VAS, where 0 = no arthritis activity to 100 = extremely active arthritis.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
mm | 65.2 (24.53) | 63.3 (9.61) | 69.0 (9.00) | 64.4 (23.33) | 64.9 (22.30)

5. Primary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Scores at Baseline
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related quality of life. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question is evaluated according to the degree of severity on a 4-point scale. Total score for HAQ-DI is the average of all questions and ranges from 0 = without any difficulty to 3 = unable to do.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 24 | 6 | 3 | 27 | 30
units on a scale | 1.7 (0.86) | 1.7 (0.98) | 1.7 (0.59) | 1.7 (0.90) | 1.7 (0.87)

6. Primary Outcome: Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Baseline
Description: TJC was determined by examining 28 and 68 joints and identifying the joints that were painful under pressure or to passive motion. Tenderness was recorded on the joint assessment form at baseline, no tenderness = 0, tenderness = 1. SJC was determined by examining 28 and 66 joints and identifying when swelling was present. Swelling was recorded on the joint assessment form at baseline, no swelling = 0, swelling =1.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with available data for the specified category.
Measure: Mean (Standard Deviation); unit: joint counts
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 27 | 6 | 4 | 29 | 33
joint counts
  TJC28 (n= 27, 6, 4, 29, 33) | 15.6 (7.68) | 14.7 (8.48) | 13.0 (8.41) | 15.8 (7.69) | 15.4 (7.70)
  TJC68 (n= 18, 5, 2, 21, 23) | 34.4 (16.97) | 24.2 (18.43) | 26.0 (7.07) | 32.8 (18.07) | 32.2 (17.40)
  SJC28 (n= 27, 6, 4, 29, 33) | 14.0 (6.66) | 14.0 (7.51) | 12.5 (3.79) | 14.2 (7.03) | 14.0 (6.70)
  SJC66 (n= 18, 5, 2, 21, 23) | 27.7 (13.73) | 21.0 (13.62) | 26.5 (7.78) | 26.2 (14.25) | 26.3 (13.69)

7. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Baseline
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeters per hour (mm/hr). A decrease in the level indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 6 | 5 | 30 | 35
mm/hr | 27.0 (24.79) | 35.2 (36.78) | 34.8 (26.79) | 27.3 (27.04) | 28.4 (26.74)

8. Primary Outcome: C-Reactive Protein (CRP) at Baseline
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline
Population: FAS population.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
milligrams per liter (mg/L) | 15.3 (17.36) | 22.6 (42.91) | 22.5 (24.30) | 16.0 (24.84) | 16.9 (24.53)

9. Secondary Outcome: Percentage of Participants Starting Tocilizumab After Stopping a Biologic Treatment or After Failing DMARDs
Time Frame: Baseline
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
percentage of participants
  Previous biologic therapy | 0 | 100 | 40 | 18.8 | 21.6
  Previous DMARD therapy | 31.0 | 7.5 | 100 | 34.4 | 43.2

10. Secondary Outcome: Median Dose at Month 6
Time Frame: Month 6
Population: FAS population. Here Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Median (Full Range); unit: milligram per kilogram (mg/kg)
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 23 | 8 | 4 | 27 | 31
milligram per kilogram (mg/kg) | 8 [7 to 8] | 8 [8 to 8] | 8 [8 to 8] | 8 [7 to 8] | 8 [7 to 8]

11. Secondary Outcome: Percentage of Participants With Tocilizumab Dose Changed According to the Reason for Change
Description: Percentage of participants with increase or decrease in tocilizumab administration according to the reason for dose modification was reported.
Time Frame: Baseline up to Month 6
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
percentage of participants
  Increase in dose | 0 | 12.5 | 0 | 3.1 | 2.7
  Decrease in dose | 3.4 | 0 | 0 | 3.1 | 2.7
  Reason:Unspecified | 3.4 | 12.5 | 0 | 6.3 | 5.4

12. Secondary Outcome: Mean Dosing Interval at Month 6
Description: The time interval between two successive doses in days was reported.
Time Frame: Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 28 | 8 | 5 | 31 | 36
days | 30.97 (3.803) | 32.10 (3.783) | 29.63 (1.505) | 31.48 (3.978) | 31.22 (3.775)

13. Secondary Outcome: Percentage of Participants With Reasons Who Discontinued Tocilizumab
Time Frame: Baseline up to Month 6
Population: FAS population. Here, Number of Participants Analyzed (N) signifies participants who discontinued tocilizumab treatment.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 5 | 0 | 1 | 4 | 5
percentage of participants
  Lack of efficacy | 20.0 |  | 0 | 25.0 | 20.0
  Adverse event | 40.0 |  | 0 | 50.0 | 40.0
  Unspecified | 40.0 |  | 100.0 | 25.0 | 40.0

14. Secondary Outcome: Time to Restoration of Initial Dosing Regimen
Time Frame: Baseline up to Month 6
Population: Analysis was not performed due to inadequate data available for this outcome measure.
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants by Reason for Choice of Monotherapy at Baseline
Time Frame: Baseline up to Month 6
Population: Analysis was not performed as the data was not collected on case report form.
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants on Tocilizumab Monotherapy (8 mg/Kg) at Baseline and at Month 6
Time Frame: Baseline, Month 6
Population: FAS population. n= participants with available data at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
percentage of participants
  Baseline (n=29,8,5,32,37) | 93.1 | 100 | 100.0 | 93.8 | 94.6
  Month 6 (n=20,8,4,24,28) | 87.0 | 100 | 100.0 | 88.9 | 90.3

17. Secondary Outcome: Duration of Tocilizumab Treatment
Time Frame: Baseline up to Month 6
Population: FAS population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
days | 181.1 (56.31) | 211.3 (28.17) | 174.8 (48.43) | 189.7 (53.79) | 187.6 (52.71)

18. Secondary Outcome: Percentage of Participants by Duration of Morning Stiffness
Description: Duration of morning stiffness was defined as the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant assessment of morning stiffness was measured using a ruler on a 100 mm VAS by 1 of the six categories: less than (<) 30 minutes, between 30 and 240 minutes, greater than (>) 240 minutes and whole day.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, n= participants with available data at specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 29 | 8 | 5 | 32 | 37
percentage of participants
  Baseline ( < 30 minutes) (n= 22, 6, 2, 26, 28) | 4.5 | 16.7 | 0 | 7.7 | 7.1
  Month 3 (< 30 minutes) (n=13, 4, 3, 14, 17) | 30.8 | 75.0 | 33.3 | 42.9 | 41.2
  Month 6 (< 30 minutes) (n= 12, 3, 3, 12, 15) | 33.3 | 0 | 0 | 33.3 | 26.7
  Baseline (30-60 minutes) (n= 22, 6, 2, 26, 28) | 13.6 | 16.7 | 0 | 15.4 | 14.3
  Month 3 (30-60 minutes) (n= 13, 4, 3, 14, 17) | 53.8 | 0 | 33.3 | 42.9 | 41.2
  Month 6 (30-60 minutes) (n= 12, 3, 3, 12, 15) | 16.7 | 66.7 | 66.7 | 16.7 | 26.7
  Baseline (60-120 minutes) (n= 22, 6, 2, 26, 28) | 18.2 | 16.7 | 50.0 | 15.4 | 17.9
  Month 3 (60-120 minutes) (n= 13, 4, 3, 14, 17) | 7.7 | 25.0 | 33.3 | 7.1 | 11.8
  Month 6 (60-120 minutes) (n= 12, 3, 3, 12, 15) | 8.3 | 0 | 0 | 8.3 | 6.7
  Baseline (120-240 minutes) (n= 22, 6, 2, 26, 28) | 31.8 | 33.3 | 0 | 34.6 | 32.1
  Month 3 (120-240 minutes) (n= 13, 4, 3, 14, 17) | 0 | 0 | 0 | 0 | 0
  Month 6 (120-240 minutes) (n=12, 3, 3, 12, 15) | 25.0 | 0 | 0 | 25.0 | 20.0
  Baseline (> 240 minutes) (n= 22, 6, 2, 26, 28) | 22.7 | 16.7 | 50.0 | 19.2 | 21.4
  Month 3 (> 240 minutes) (n= 13, 4, 3, 14, 17) | 0 | 0 | 0 | 0 | 0
  Month 6 (> 240 minutes) (n= 12, 3, 3, 12, 15) | 8.3 | 33.3 | 33.3 | 8.3 | 13.3
  Baseline (whole day) (n= 22, 6, 2, 26, 28) | 9.1 | 0 | 0 | 7.7 | 7.1
  Month 3 (whole day) (n= 13, 4, 3, 14, 17) | 7.7 | 0 | 0 | 7.1 | 5.9
  Month 6 (whole day) (n= 12, 3, 3, 12, 15) | 8.3 | 0 | 0 | 8.3 | 6.7

19. Secondary Outcome: Percentage of Participants With and Without Morning Stiffness
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. The participant assessed morning stiffness based on the following criteria:
  1. Presence of participant's joints stiff when woke up that day, measured as yes or no
  2. Duration of morning stiffness, measured using a ruler on a 100 mm VAS by 1 of the six categories: < 30 minutes, between 30 and 240 minutes, > 240 minutes, and the whole day.
  3. Severity of morning stiffness measured using a ruler on a 100 mm VAS where the responses were on a continuous range from 0 = no stiffness to 100 = maximum stiffness.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with available data at the specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 24 | 6 | 4 | 27 | 30
percentage of participants
  Baseline(with morning stiffness)(n=24,6,3,27,30) | 95.8 | 100 | 100 | 96.3 | 96.7
  Baseline(without morningstiffness)(n=24,6,3,27,30) | 4.2 | 0 | 0 | 3.7 | 3.3
  Month 3(with morning stiffness)(n=14,5,4,15,19) | 92.9 | 100 | 100 | 93.3 | 94.7
  Month 3(without morning stiffness)(n=14,5,4,15,19) | 7.1 | 0 | 0 | 6.7 | 5.3
  Month 6(with morning stiffness)(n=14,3,4,13,17) | 92.9 | 100 | 100 | 92.3 | 94.1
  Month 6(without morning stiffness)(n=14,3,4,13,17) | 17.1 | 0 | 0 | 7.7 | 5.9

20. Secondary Outcome: Percentage of Participants Adhering to Local Label for Adverse Events
Description: Percentage of participants who adhered to local label/protocol for the management of adverse events is reported.
Time Frame: Baseline up to Month 6
Population: FAS population. Number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 4 | 1 | 1 | 4 | 5
percentage of participants | 100 | 100 | 100 | 75 | 80

21. Secondary Outcome: Disease Activity Score Based on 28 Joint Count (DAS28) Score by Visit
Description: The DAS28 score is a measurement of RA activity on a 0 to 10 scale, with higher scores representing higher disease activity, and calculated as DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.70 x natural logarithm (ln) (CRP + 1) + 0.014 x PGH + 0.96, where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, CRP = serum concentration of c-reactive protein (after converting units to mg/dL), PGH = patient global assessment of disease activity, which was measured on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly. A score of less than 2.6 represents clinical remission, a score of greater than or equal to 2.6 and less than or equal to 3.2 represents low disease activity, a score of greater than 3.2 and less than or equal to 5.1 represents moderate disease activity, and a score of greater than 5.1 represents high (or severe) disease.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = Participants evaluable for the outcome measure and n= participants with DAS28 score available at the specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 22 | 6 | 3 | 25 | 28
units on a scale
  Baseline (n=22, 6, 3, 25, 28) | 6.34 (1.611) | 6.04 (1.272) | 6.73 (0.868) | 6.22 (1.592) | 6.28 (1.528)
  Month 3 (n=13, 4, 2, 15, 17) | 2.69 (1.274) | 2.98 (1.250) | 3.61 (0.151) | 2.64 (1.275) | 2.76 (1.236)
  Month 6 (n=12, 2, 2, 12, 14) | 3.02 (1.459) | 2.75 (1.420) | 3.49 (0.380) | 2.89 (1.502) | 2.98 (1.402)

22. Secondary Outcome: Percentage of Participants Achieving Good European League Against Rheumatism (EULAR) Response at Month 3 and Month 6
Description: Clinical response was assessed according to EULAR criteria that classified the participant according to individual changes in DAS28 score as good, moderate, or no response. The DAS28 score is a measurement of RA activity on a 0 to 10 scale, with higher scores represent higher disease activity, and calculated as DAS28 = 0.56 x √TJC28 + 0.28 x √SJC28 + 0.36 x ln(CRP + 1) + 0.014 x PGH + 0.96, where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, CRP = serum concentration of c-reactive protein (after converting units to mg/dL), PGH = patient's global assessment of disease activity, which was measured on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly. Good responders experienced a change from baseline of greater than 1.2 with a DAS28 score less than or equal to 3.2.
Time Frame: Month 3 and Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with EULAR response available at specified visit.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 11 | 3 | 1 | 13 | 14
percentage of participants
  Month 3 (n= 11, 3, 1, 13, 14) | 63.6 | 66.7 | 0 | 69.2 | 64.3
  Month 6 (n= 10, 1,1, 10, 11) | 50.0 | 100 | 0 | 60.0 | 54.5

23. Secondary Outcome: Clinical Disease Activity Index (CDAI) Score by Visit
Description: The CDAI is a combined index for measuring disease activity in RA and calculated as CDAI = TJC28 + SJC28 + PGH (in centimeters) + PhGH (in centimeters), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly, and PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 = no arthritis activity and 100 = extremely active arthritis; with a total score ranged from 0-76. Higher scores indicate greater disease activity. CDAI score of less than or equal to 2.8 represents clinical remission, score of less than or equal to 10.0 represents low disease activity, score of less than or equal to 22.0 represents moderate disease activity, and score of greater than 22.0 represents high (or severe) disease.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with CDAI score available at specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 22 | 6 | 4 | 25 | 28
units on a scale
  Baseline (n= 22, 6, 3, 25, 28) | 46.41 (16.482) | 40.90 (18.277) | 45.40 (4.900) | 45.21 (17.643) | 45.23 (16.687)
  Month 3 (n= 13, 5, 4, 14, 18) | 12.37 (10.970) | 16.00 (5.632) | 13.05 (7.468) | 13.47 (10.564) | 13.38 (9.758)
  Month 6 (n= 13, 3, 4, 12, 16) | 13.20 (15.017) | 14.93 (4.140) | 11.30 (7.338) | 14.27 (15.254) | 13.53 (13.534)

24. Secondary Outcome: Change From Baseline in TJC and SJC at Month 3 and Month 6
Description: TJC was determined by examining 28 and 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at baseline, no tenderness = 0, tenderness = 1. SJC was determined by examination of 28 and 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at baseline, no swelling = 0, swelling =1.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: joint counts
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 27 | 6 | 4 | 29 | 33
joint counts
  TJC28: Baseline (n= 27, 6, 4, 29, 33) | 15.6 (7.68) | 14.7 (8.48) | 13.0 (8.41) | 15.8 (7.69) | 15.4 (7.70)
  TJC28: Change at Month 3 (n= 14, 4, 3, 15, 18) | -13.9 (5.17) | -11.0 (6.78) | -7.0 (5.57) | -14.5 (4.70) | -13.2 (5.48)
  TJC28: Change at Month 6 (n= 14, 2, 3, 13, 16) | -11.1 (8.56) | -15.0 (7.07) | -8.3 (6.66) | -12.3 (8.67) | -11.6 (8.29)
  TJC68: Baseline (n= 18, 5, 2, 21, 23 ) | 34.4 (16.97) | 24.2 (18.43) | 26.0 (7.07) | 32.8 (18.07) | 32.2 (17.40)
  TJC68: Change at Month 3 (n= 11, 3, 2, 12, 14) | -30.5 (8.13) | -12.3 (6.66) | -18.0 (12.73) | -28.1 (10.42) | -26.6 (10.85)
  TJC68: Change at Month 6 (n= 11, 1, 2, 10, 12 ) | -27.5 (17.41) | -17.0 (NA) — SD not calculable because only 1 participant was evaluated. | -21.5 (6.36) | -27.7 (18.34) | -26.7 (16.88)
  SJC28: Baseline (n= 27, 6, 4, 29, 33) | 14.0 (6.66) | 14.0 (7.51) | 12.5 (3.79) | 14.2 (7.03) | 14.0 (6.70)
  SJC28: Change at Month 3 (n= 14, 4, 3, 15, 18) | -13.8 (4.54) | -10.5 (6.81) | -9.3 (5.51) | -13.8 (4.86) | -13.1 (5.09)
  SJC28: Change at Month 6 (n= 14, 2, 3, 13, 16) | -10.8 (6.34) | -13.5 (4.95) | -11.7 (2.89) | -11.0 (6.72) | -11.1 (6.11)
  SJC66: Baseline (n= 18, 5, 2, 21, 23) | 27.7 (13.73) | 21.0 (13.62) | 26.5 (7.78) | 26.2 (14.25) | 26.3 (13.69)
  SJC66: Change at Month 3 (n= 11, 3, 2, 12, 14) | -27.2 (9.58) | -12.7 (5.51) | -18.5 (13.44) | -25.0 (10.54) | -24.1 (10.65)
  SJC66: Change at Month 6 (n= 11, 1, 2, 10, 12) | -26.0 (13.80) | -17.0 (NA) — SD not calculable because only 1 participant was evaluated. | -21.5 (6.36) | -26.0 (14.54) | -25.3 (13.41)

25. Secondary Outcome: Simplified Disease Activity Index (SDAI) Score by Visit
Description: The SDAI is a combined index for measuring disease activity in RA and calculated as SDAI = TJC28 + SJC28 + PGH (in centimeters) + PhGH (in centimeters) + CRP (in mg/dL), where TJC28 = tender joint count on 28 units, SJC28 = swollen joint count on 28 units, PGH = patient's global assessment of disease activity, assessed on a 100 mm VAS, where 0 = managing very well and 100 = managing very poorly, PhGH = physician global assessment of disease activity, assessed on a 100 mm VAS, where 0 = no arthritis activity and 100 = extremely active arthritis, CRP = serum concentration of c-reactive protein; with a total SDAI score ranged from 0-86. Higher scores indicate greater disease activity. SDAI scores of less than or equal to 3.3 represents clinical remission, less than or equal to 11.0 represents low disease activity, less than or equal to 26.0 represents moderate disease activity, and greater than 26.0 represents high (or severe) disease.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with SDAI score available at the specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 22 | 6 | 3 | 25 | 28
units on a scale
  Baseline (n= 22, 6, 3, 25, 28) | 48.01 (16.853) | 43.57 (14.898) | 47.07 (6.689) | 47.06 (17.173) | 47.06 (16.293)
  Month 3 (n= 11, 4, 2, 13, 15) | 13.29 (11.602) | 15.16 (6.066) | 14.95 (3.536) | 13.61 (10.997) | 13.79 (10.236)
  Month 6 (n= 12, 2, 2, 12, 14) | 14.55 (15.357) | 14.65 (5.798) | 13.70 (7.142) | 14.70 (15.301) | 14.56 (14.218)

26. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20%, 50%, or 70% (ACR20/50/70) Response at Month 3 and Month 6 From the Start of Tocilizumab Treatment
Description: ACR 20,50 or 70 response=an improvement of ≥ 20%, ≥ 50% or ≥ 70% respectively, as compared to baseline in TJC28 and SJC28, and 20%, 50% or 70% improvement in at least 3 of the 5 following measures: Patient's Assessment of Pain over the previous 24 hours, PGA, PhGA, HAQ, and acute phase reactant (either CRP or ESR). TJC and SJC, based on 28-joint assessments. Number of tender joints and swollen joints were recorded on the joint assessment form at baseline, no tenderness = 0 and tenderness = 1, no swelling = 0 and swelling =1, respectively. HAQ measures functional status (disability) and health-related quality of life with 20 questions, summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week, 0=without difficulty to 3=unable to do. Patient's assessment of pain assessed using a VAS; 0=no pain, 100=unbearable pain; PGA and PhGA, assessed using VAS ; 0= no disease activity, 100=maximum disease activity.
Time Frame: Month 3 and Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n= participants with available data for the specified visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 11 | 3 | 2 | 12 | 14
percentage of participants
  Month 3: ACR20 responders (n= 11, 3, 2, 12, 14) | 90.9 [58.7 to 99.8] | 100.0 [29.2 to 100] | 100.0 [15.8 to 100] | 91.7 [61.5 to 99.8] | 92.9 [66.1 to 99.8]
  Month 6: ACR20 responders (n= 10, 1, 2, 9, 11) | 80.0 [44.4 to 97.5] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100] | 77.8 [40.0 to 97.2] | 81.8 [48.2 to 97.7]
  Month 3: ACR50 responders (n= 11, 3, 2, 12, 14) | 63.6 [30.8 to 89.1] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 84.2] | 66.7 [34.9 to 90.1] | 57.1 [28.9 to 82.3]
  Month 6: ACR50 responders (n= 10, 1, 2, 9, 11) | 70.0 [34.8 to 93.3] | 0.0 [0.0 to 97.5] | 50.0 [1.3 to 98.7] | 66.7 [29.9 to 92.5] | 63.6 [30.8 to 89.1]
  Month 3: ACR70 responders (n= 11, 3, 2, 12, 14) | 36.4 [10.9 to 69.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 33.3 [9.9 to 65.1] | 28.6 [8.4 to 58.1]
  Month 6: ACR70 responders (n= 10, 1, 2, 9, 11) | 50.0 [18.7 to 81.3] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2] | 55.6 [21.2 to 86.3] | 45.5 [16.7 to 76.6]

27. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Months 3 and 6
Description: The physician global assessment of disease activity was evaluated using a 100 mm VAS where 0 = no arthritis activity and 100 = extremely active arthritis. Higher scores indicated increased level of disease.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
mm
  Baseline (n= 25, 6, 3, 28, 31) | 65.2 (24.53) | 63.3 (9.61) | 69.0 (9.00) | 64.4 (23.33) | 64.9 (22.30)
  Change at Month 3 (n= 13, 4, 2, 15, 17) | -40.8 (24.07) | -33.8 (11.56) | -43.5 (4.95) | -38.6 (23.05) | -39.2 (21.66)
  Change at Month 6 (n= 13, 2, 2, 13, 15) | -35.2 (28.12) | -38.5 (13.44) | -45.5 (23.33) | -34.2 (27.27) | -35.7 (26.31)

28. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity at Months 3 and 6
Description: The patient's global assessment of disease activity was measured using a 100 mm VAS, where the responses were on a continuous range from 0= managing very well and 100 = managing very poorly.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 24 | 6 | 3 | 27 | 30
mm
  Baseline (n=24, 6, 3, 27, 30) | 69.6 (29.71) | 59.0 (33.03) | 85.0 (11.36) | 65.5 (31.02) | 67.5 (30.11)
  Change at Month 3 (n= 16, 4, 2, 18, 20 ) | -43.2 (35.87) | -34.5 (18.70) | -50.0 (16.97) | -40.5 (34.42) | -41.5 (32.92)
  Change at Month 6 (n= 13, 2, 2, 13, 15) | -26.4 (31.28) | -37.0 (33.94) | -32.0 (26.87) | -27.2 (32.05) | -27.8 (30.57)

29. Secondary Outcome: Change From Baseline in HAQ-DI Score at Months 3 and 6
Description: The HAQ-DI is a questionnaire that measures functional status (disability) and health-related quality of life. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities over past week. Each question was evaluated according to the degree of severity on a 4-point scale ranging from 0 = without any difficulty to 3 = unable to do. Total score is the sum of each question, which ranges from 0 to 60, where higher scores represent higher disease activity. The change from baseline in HAQ-DI score at Month 3 and Month 6 was calculated as the difference between HAQ-D1 score reported at baseline and the HAQ-D1 score reported at Month 3 and Month 6.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n = participants with available HAQ-DI score at specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 24 | 6 | 3 | 27 | 30
units on a scale
  Baseline (n= 24, 6, 3, 27, 30) | 1.7 (0.86) | 1.7 (0.98) | 1.7 (0.59) | 1.7 (0.90) | 1.7 (0.87)
  Change at Month 3 (n= 16, 4, 2, 18, 20) | -0.5 (0.94) | -0.4 (0.37) | -0.3 (0.35) | -0.5 (0.89) | -0.5 (0.85)
  Change at Month 6 (n= 12, 2, 2, 12, 14) | -0.3 (0.48) | -0.6 (0.35) | -0.4 (0.09) | -0.3 (0.51) | -0.3 (0.46)

30. Secondary Outcome: Change From Baseline in VAS-Fatigue at Months 3 and 6
Description: Participants measured the level of fatigue due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 = no fatigue to 100 = extreme fatigue.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
mm
  Baseline (n= 25, 6, 3, 28, 31) | 59.0 (34.35) | 67.8 (27.01) | 86.3 (8.08) | 58.0 (33.35) | 60.7 (32.84)
  Change at Month 3 (n= 16, 4, 2, 18, 20) | -23.2 (29.90) | -37.8 (24.93) | -38.5 (13.44) | -24.7 (30.13) | -26.1 (28.98)
  Change at Month 6 (n=12, 2, 2, 12, 14) | -19.8 (29.81) | -34.0 (22.63) | -51.5 (2.12) | -16.8 (27.91) | -21.8 (28.60)

31. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Months 3 and 6
Description: Participants measured the pain intensity due to RA using a 100 mm VAS, where the responses were on a continuous range from 0 = no pain to 100 = unbearable pain.
Time Frame: Baseline, Month 3, Month 6
Population: FAS population. Here, Number of participants analyzed = participants evaluable for the outcome measure and n = participants with available data for the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
mm
  Baseline (n= 25, 6, 3, 28, 31) | 60.1 (31.08) | 47.2 (31.93) | 79.3 (19.55) | 55.3 (31.49) | 57.6 (31.14)
  Change at Month 3 (n= 16, 4, 2, 18, 20) | -35.6 (39.39) | -15.8 (26.99) | -39.5 (14.85) | -30.8 (39.38) | -31.17 (37.50)
  Change at Month 6 (n= 13, 2, 2, 13, 15) | -32.3 (34.88) | -47.0 (14.14) | -51.5 (7.78) | -31.6 (34.68) | -34.3 (32.93)

32. Secondary Outcome: Change From Baseline in Participant Assessment of Morning Stiffness Using VAS at Months 3 and 6
Description: The participant assessment of morning stiffness was measured using a ruler on a 100 mm VAS, where the responses were on a continuous range from 0 = no stiffness and 100 = maximum stiffness.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RA Participants (Biologic Naïve Group) | RA Participants (Biologic Exposed Group) | RA Participants (Monotherapy Group) | RA Participants (Combination Therapy Group) | RA Participants (All Groups)
Number analyzed (Participants) | 25 | 6 | 3 | 28 | 31
mm
  Baseline (n= 25, 6, 3, 28, 31) | 65.6 (31.29) | 57.3 (29.92) | 77.3 (22.03) | 62.5 (31.46) | 64.0 (30.71)
  Change at Month 3 (n= 15, 4, 2, 17, 19) | -30.7 (37.88) | -34.0 (17.80) | -42.5 (14.85) | -30.1 (35.86) | -31.4 (34.21)
  Change at Month 6 (n= 12, 2, 2, 12, 14) | -30.2 (35.88) | -38.0 (14.14) | -31.5 (4.95) | -31.3 (36.23) | -31.3 (33.35)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from enrollment up to 6 months (final visit).
Arm/Group | RA Participants (All Groups)
Serious Adverse Events (participants affected / at risk) | 2/37
Other Adverse Events (participants affected / at risk) | 12/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA Participants (All Groups) (N=37)
Mycoplasma infection (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RA Participants (All Groups) (N=37)
Neutropenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.